CLINICAL TRIAL: NCT04330690
Title: A Multi-centre, Adaptive, Randomized, Open-label, Controlled Clinical Trial of the Safety and Efficacy of Investigational Therapeutics for the Treatment of COVID-19 in Hospitalized Patients (CATCO: Canadian Treatments for COVID-19), in Conjunction With the Public Health Emergency SOLIDARITY Trial (World Health Organization)
Brief Title: Treatments for COVID-19: Canadian Arm of the SOLIDARITY Trial
Acronym: CATCO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: AbbVie (Industry); Apotex Inc. (Industry); World Health Organization (Other); University of British Columbia (Other); Arch Biopartners Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2114
Record Dates: First submitted 2020-03-23; First posted 2020-04-01 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: Artesunate; Infliximab; Imatinib; Dexamethasone; SARS-CoV-2; LSALT Peptide
MeSH Terms: conditions — COVID-19 | interventions — Artesunate; Imatinib Mesylate; Infliximab; Dexamethasone

STUDY DESIGN:
Masking Description: Endpoint assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Artesunate (Experimental): Subjects will be randomized Artesunate vs Imatinib vs Infliximab vs standard of care
  Interventions: Drug: Artesunate
- Imatinib (Experimental): Subjects will be randomized Artesunate vs Imatinib vs Infliximab vs standard of care
  Interventions: Drug: Imatinib
- Infliximab (Experimental): Subjects will be randomized Artesunate vs Imatinib vs Infliximab vs standard of care
  Interventions: Drug: Infliximab
- Dexamethasone (Experimental): Subjects will be randomized between Dexamethasone vs standard of care.
  Interventions: Drug: Dexamethasone
- LSALT Peptide (Experimental): Subjects will be randomized between LSALT vs standard of care.
  Interventions: Drug: LSALT Peptide
- Control (Standard Care) (No Intervention): This arm will receive standard supportive care guidelines for COVID-19. It is expected to vary regionally and may change throughout the trial based on new and emerging data on best care guidelines for patients.

INTERVENTIONS:
Drug: Artesunate — 2.4 mg/kg at 0 hours, 12 hours, 24 hours, and then daily for a total of 7 days plus standard of care
  Arms: Artesunate
Drug: Imatinib — 400 mg enterally daily for 14 days plus standard of care
  Arms: Imatinib
Drug: Infliximab — 5 mg/kg IV given one time, over 2 hours plus standard of care
  Arms: Infliximab
Drug: Dexamethasone — 6 mg IV/oral for a further five days, followed by a five day taper of 4 mg x 2 days and 2 mg x 3 days, for a total 20 day steroid course. If randomized to standard of care, discontinue the corticosteroid on day 10
  Arms: Dexamethasone
Drug: LSALT Peptide — 5 mg , 2 hour IV infusion once daily for up to 14 consecutive days
  Arms: LSALT Peptide

SUMMARY:
This study is an adaptive, randomized, open-label, controlled clinical trial, in collaboration with countries around the world through the World Health Organization.

DETAILED DESCRIPTION:
Subjects will be randomized, across one, two, three or up to four separate randomizations, to receive either standard-of-care products or the study medication plus standard of care, while being hospitalized for COVID-19.

Randomization WHO: Imatinib vs Infliximab vs Artesunate vs Standard of care

Randomization Dex: Dexamethasone vs Standard of care

Randomization LSALT: LSALT Peptide vs Standard of care

Hospitalized subjects will require blood sampling for screening and on days 1 and 5.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria to participate in this study:

1. ≥ 18 years of age
2. Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen, within 14 days prior to randomization.
3. Hospitalized at a participating centre
4. Primary reason for hospitalization or subsequent in-hospital illness is because of acute COVID19 infection
5. First admission for acute COVID19

In addition, there will be the below intervention-specific inclusion:

Randomization WHO will have no other specific inclusion criteria.

Randomization LSALT will have no other specific inclusion criteria.

Randomization Dex will have the following specific inclusion criteria

1. On 10 days of steroid course and
2. Receiving any supplemental oxygen for 10 days

Exclusion Criteria:

All participants meeting any of the following exclusion criteria at baseline will be excluded from participation in this study:

1. Anticipated transfer to another hospital, within 72 hours, which is not a study site
2. Expected to not survive beyond 24 hours
3. Receiving one of the study drugs at time of enrolment

In addition, there will be the below intervention-specific exclusions:

Randomization WHO:

These will be drug-specific exclusions; patients will still be eligible for randomization in Randomization WHO to the other available study drugs (in randomization WHO or subsequent randomizations).

Artesunate:

1. Known hypersensitivity to artesunate

Imatinib:

1. Pregnant or breastfeeding;
2. Known hypersensitivity to imatinib;
3. Liver transaminases (either ALT or AST) > 5x upper limit of normal

Infliximab:

1. Known moderate or severe heart failure, per treating clinician, defined as New York Heart Association (NYHA) class III or IV
2. Known or suspected active tuberculosis
3. Known hypersensitivity to infliximab

Randomization LSALT:

1. Known hypersensitivity or prior use of LSALT peptide.
2. Pregnant or breastfeeding

Randomization Dex:

1. Receiving glucocorticoids for a specific, non-COVID-19 indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2900 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-05-18 (Estimated)

PRIMARY OUTCOMES:
Randomization WHO- Mortality | 28 days
  All-cause mortality, assessed at hospital discharge.
Randomization Dex- Clinical Status | 28 days
  Position on the WHO Ordinal scale at 28 days post-randomization.
  Ordinal Scale Table:
  0 Uninfected; 1-3 Ambulatory; 4-5 Hospitalized/ Mild disease; 6-9 Hospitalized/ Severe Disease; 10 Death
Randomization LSALT- Respiratory support | 28 days
  Number of days respiratory support free days

SECONDARY OUTCOMES:
Evaluation of the clinical effectiveness of study drugs | 24 months
  To be compared to the control arm on duration of hospitalization
Need for invasive mechanical ventilation | 24 months
CU admission, hospital and ICU length of stay, days alive and free of vasopressors, ventilation, and renal replacement therapy (RRT | 24 months
Mortality | 12 months
  Mortality after Randomization

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Murthy, MD, Principal Investigator — Provincial Health Services Authority British Columbia
Locations (53):
- Canada (53):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - University of Alberta Hopsital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Interior Health Royal Inland Hospital, Kamloops, British Columbia
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Richmond Hospital, Richmond, British Columbia
  - Vancouver General Hospital, Vancouver Coastal Health, Univeristy of British Columbia, Vancouver, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia
  - Island Health - Royal Jubilee Hospital, Victoria, British Columbia
  - Island Health - Victoria General Hospital, Victoria, British Columbia
  - Island Health - Nanaimo Regional General Hospital, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - Grace General Hospital, Winnipeg, Manitoba
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Health System - Brampton Civic Hospital, Brampton, Ontario
  - William Osler Health System - Etobicoke General Hospital, Etobicoke, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - St.Joseph's Health Care, London, Ontario
  - University Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Trillium Health Partners -Mississauga Site, Mississauga, Ontario
  - Trillium Health Partners-Credit Valley Hospital, Mississauga, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Hôpital Montfort, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Queensway Carleton Hospital, Ottawa, Ontario
  - Niagara Health, Saint Catharines, Ontario
  - Scarborough Health Network - Centenary Hospital, Scarborough Village, Ontario
  - Scarborough Health Network - General Hospital, Scarborough Village, Ontario
  - Scarborough Health Network - Birchmount Hospital, Scarborough Village, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - North York General Hospital, Toronto, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Unity Health Toronto - St. Joseph's Health Centre, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - McGill University Health Centre-Glen Site Royal Victoria Hospital, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec- Université Laval, Québec, Quebec
  - Centre Intégré Universitaire de Santé et de Services Sociaux de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
As per World Health Organization policies on data sharing in a Public Health Emergency, any clinical trial outcome data will be shared at the earliest possible opportunity. In addition, given the nature of this protocol, being performed across regions, the DSMB may access other regions trials, and possibly recommend alterations in study design based on accumulating data, through a centralized data repository being built under the auspices of the World Health Organization.
  Data Sharing for Secondary Research Data from this study may be used for secondary research. All of the individual subject data collected during the trial will be made available after de-identification through expert determination. The SAP and Analytic Code will also be made available. This data will be available immediately following publication, with no end date, as part of data sharing requirements from journals and funding agencies.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Unknown and variable

REFERENCES:
- [Result] Ali K, Azher T, Baqi M, Binnie A, Borgia S, Carrier FM, Cavayas YA, Chagnon N, Cheng MP, Conly J, Costiniuk C, Daley P, Daneman N, Douglas J, Downey C, Duan E, Duceppe E, Durand M, English S, Farjou G, Fera E, Fontela P, Fowler R, Fralick M, Geagea A, Grant J, Harrison LB, Havey T, Hoang H, Kelly LE, Keynan Y, Khwaja K, Klein G, Klein M, Kolan C, Kronfli N, Lamontagne F, Lau R, Fralick M, Lee TC, Lee N, Lim R, Longo S, Lostun A, MacIntyre E, Malhame I, Mangof K, McGuinty M, Mergler S, Munan MP, Murthy S, O'Neil C, Ovakim D, Papenburg J, Parhar K, Parvathy SN, Patel C, Perez-Patrigeon S, Pinto R, Rajakumaran S, Rishu A, Roba-Oshin M, Rushton M, Saleem M, Salvadori M, Scherr K, Schwartz K, Semret M, Silverman M, Singh A, Sligl W, Smith S, Somayaji R, Tan DHS, Tobin S, Todd M, Tran TV, Tremblay A, Tsang J, Turgeon A, Vakil E, Weatherald J, Yansouni C, Zarychanski R; Canadian Treatments for COVID-19 (CATCO); Association of Medical Microbiology and Infectious Disease Canada (AMMI) Clinical Research Network and the Canadian Critical Care Trials Group. Remdesivir for the treatment of patients in hospital with COVID-19 in Canada: a randomized controlled trial. CMAJ. 2022 Feb 22;194(7):E242-E251. doi: 10.1503/cmaj.211698. Epub 2022 Jan 19. PMID 35045989
- [Result] WHO Solidarity Trial Consortium; Pan H, Peto R, Henao-Restrepo AM, Preziosi MP, Sathiyamoorthy V, Abdool Karim Q, Alejandria MM, Hernandez Garcia C, Kieny MP, Malekzadeh R, Murthy S, Reddy KS, Roses Periago M, Abi Hanna P, Ader F, Al-Bader AM, Alhasawi A, Allum E, Alotaibi A, Alvarez-Moreno CA, Appadoo S, Asiri A, Aukrust P, Barratt-Due A, Bellani S, Branca M, Cappel-Porter HBC, Cerrato N, Chow TS, Como N, Eustace J, Garcia PJ, Godbole S, Gotuzzo E, Griskevicius L, Hamra R, Hassan M, Hassany M, Hutton D, Irmansyah I, Jancoriene L, Kirwan J, Kumar S, Lennon P, Lopardo G, Lydon P, Magrini N, Maguire T, Manevska S, Manuel O, McGinty S, Medina MT, Mesa Rubio ML, Miranda-Montoya MC, Nel J, Nunes EP, Perola M, Portoles A, Rasmin MR, Raza A, Rees H, Reges PPS, Rogers CA, Salami K, Salvadori MI, Sinani N, Sterne JAC, Stevanovikj M, Tacconelli E, Tikkinen KAO, Trelle S, Zaid H, Rottingen JA, Swaminathan S. Repurposed Antiviral Drugs for Covid-19 - Interim WHO Solidarity Trial Results. N Engl J Med. 2021 Feb 11;384(6):497-511. doi: 10.1056/NEJMoa2023184. Epub 2020 Dec 2. PMID 33264556
- [Result] Cheng M, Fowler R, Murthy S, Pinto R, Sheehan NL, Tseng A. Remdesivir in Patients With Severe Kidney Dysfunction: A Secondary Analysis of the CATCO Randomized Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2229236. doi: 10.1001/jamanetworkopen.2022.29236. PMID 36036936
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- [Derived] Lau VI, Fowler R, Pinto R, Tremblay A, Borgia S, Carrier FM, Cheng MP, Conly J, Costiniuk CT, Daley P, Duan E, Durand M, Fontela PS, Farjou G, Fralick M, Geagea A, Grant J, Keynan Y, Khwaja K, Lee N, Lee TC, Lim R, O'Neil CR, Papenburg J, Semret M, Silverman M, Sligl W, Somayaji R, Tan DHS, Tsang JLY, Weatherald J, Yansouni CP, Zarychanski R, Murthy S; E-CATCO authors, AMMI Clinical Research Network and Canadian Critical Care Trials Group. Cost-effectiveness of remdesivir plus usual care versus usual care alone for hospitalized patients with COVID-19: an economic evaluation as part of the Canadian Treatments for COVID-19 (CATCO) randomized clinical trial. CMAJ Open. 2022 Sep 6;10(3):E807-E817. doi: 10.9778/cmajo.20220077. Print 2022 Jul-Sep. PMID 36199248
- [Derived] Essai CATCO (Canadian Treatments for COVID-19); pour le Reseau de recherche clinique de l'Association pour la microbiologie medicale et l'infectiologie Canada (AMMI Canada) le Groupe canadien de recherche en soins intensifs (CCCTG). Remdesivir chez les patients hospitalises pour la COVID-19 au Canada: essai clinique randomise et controle. CMAJ. 2022 May 24;194(20):E713-E723. doi: 10.1503/cmaj.211698-f. French. PMID 35609913
- [Derived] Ansems K, Grundeis F, Dahms K, Mikolajewska A, Thieme V, Piechotta V, Metzendorf MI, Stegemann M, Benstoem C, Fichtner F. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD014962. doi: 10.1002/14651858.CD014962. PMID 34350582
- See also: Remdesivir for the treatment of patients in hospital with COVID-19 in Canada: a randomized controlled trial — https://www.cmaj.ca/content/194/7/E242
- See also: Repurposed Antiviral Drugs for Covid-19 - Interim WHO Solidarity Trial Results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7727327/